CLINICAL TRIAL: NCT03782129
Title: Five-year Mortality Rate in People With Diabetic Foot Ulcer
Acronym: DIAFOOT
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-16
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus; Diabetic Foot; Diabetes Complications
Keywords: diabetes mellitus; diabetic foot; mortality rate; diabetes complications
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients with DFU: Diabetic patients with DFU diagnosed in 2010
  Interventions: Biological: blood samples; Other: Clinical exam and DFU medical cares

INTERVENTIONS:
Biological: blood samples — Blood samples drawn during hospitalisations when needed
Other: Clinical exam and DFU medical cares — Clinical exam and DFU's medical cares at each visit (planned evry 1 to 3 months), during all the 5 years follow up, or until death.

SUMMARY:
As the global mortality rate decreases for diabetics patients, further explorations and datas are needed about the specific population of diabetics patients suffering a Diabetic Foot Ulcer (DFU).

This study investigates the 5 years mortality rate in patients with a diabetic foot ulcer occurring in 2010.

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) is an economic burden for many countries around the world. It also induces a dramatic decrease in physical, emotional, and social functioning for patients. Oftenly associated with advanced micro and macrovascular complications, high morbidity and a greater risk of premature death (mainly by Ischemic Heart Disease) occure.

Only few studies explored DFU patients' long term survival: the few datas coming from cohorts in the 2000's reported mortality rates around 45% at five years after DFU's diagnosis.

But life expectancy in diabetics patients imporved during last decade. So the main objective of our study is to evaluate the diabetics patients' 5 years mortality rate, in whom DFU was diagnosed in 2010.

Moreover, our secondary objective is to identify the mortality's predictive factors in 2010.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or 2 diabetes
* consultation for new diabetic foot ulcer during the year 2010

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with a DFU diagnosed in 2010
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mortality rate 5 years after DFU diagnosis | 5 years
  Five years after DFU diagnosis, patients are called by phone to enquire their health. If patients are dead, family tell us. If no family is available, the City Hall is called to check the death list.

SECONDARY OUTCOMES:
Risks factors correlated to mortality rate among DFU patients diagnosed in 2010 | 5 years
  All relevants staisticals associations between mortality rate and DFU diagnosed in 2010

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided